CLINICAL TRIAL: NCT06213025
Title: A Randomized Control Trials of Web-based Educational Program Promoting Response and Willingness to Handle Elderly Abuse Among Gerontological Nurses.
Brief Title: Web-based Educational Program Promoting
Acronym: web-based
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 91-c
Record Dates: First submitted 2024-01-05; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Educational Problems; Nursing Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web-based Educational program (Experimental): nurses who entered a web-based Educational program about elder abuse will demonstrate higher response and willingness to handle elderly abuse (high score in REAGERA-P scale) than those who not entered
  Interventions: Behavioral: web-based Educational program promoting response and willingness to handle elderly
- nurses in control group (No Intervention): non intervention group

INTERVENTIONS:
Behavioral: web-based Educational program promoting response and willingness to handle elderly — promote the response and willingness of gerontological nurses in handling elderly abuse cases. By employing a rigorous experimental design, this research seeks to contribute evidence-based insights that can inform educational strategies to empower nurses in safeguarding the well-being of elderly individuals.
  Arms: web-based Educational program

SUMMARY:
Elderly abuse is a pervasive and concerning issue, particularly as the global population ages. Gerontological nurses play a pivotal role in identifying, preventing, and responding to elder abuse.

DETAILED DESCRIPTION:
A virtual-based educational program designed to alter nurses' responses to violence against older adults is a comprehensive and interactive initiative aimed at equipping healthcare professionals with the knowledge, skills, and attitudes necessary to address and mitigate instances of violence within this vulnerable demographic. This program leverages digital platforms, incorporating multimedia elements, such as videos, case studies, and interactive simulations, to create an engaging and immersive learning experience. The curriculum is meticulously curated to cover various facets of violence against older adults, encompassing types of abuse, risk factors, identification strategies, and evidence-based intervention techniques.

Key components of the virtual program include scenario-based learning modules that simulate real-world situations nurses may encounter, allowing them to practice appropriate responses in a risk-free environment. Additionally, the program incorporates theoretical frameworks and ethical considerations to guide nurses in understanding the complexities of violence against older adults and formulating empathetic and effective responses.

Interactivity is a focal point, with virtual discussions, forums, and collaborative activities promoting knowledge sharing and peer learning. The program integrates assessments to measure participants' understanding and retention of the material, fostering a continuous learning process.

Moreover, the virtual program emphasizes the importance of interdisciplinary collaboration, encouraging nurses to work in tandem with other healthcare professionals, social services, and law enforcement agencies to create a comprehensive and supportive network for older adults experiencing violence.

Post-program support mechanisms, such as access to resources, expert consultations, and ongoing forums, contribute to sustaining the knowledge gained and fostering a community of practice committed to addressing violence against older adults. Overall, this virtual-based educational program serves as a dynamic and responsive platform, empowering nurses to proactively address and respond to instances of violence against older adults in a holistic and compassionate manner.

ELIGIBILITY:
Inclusion Criteria:

* willingness to enter

Exclusion Criteria:

* entered previous program about elder abuse

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
web-based educational program | three months
  nurses who entered a web-based Educational program about elder abuse will demonstrate a higher score in Responding to Elder Abuse in GERiAtric Care - Provider questionnaire to handle elderly abuse ( total score range from 15 to 75, a higher score of more than 50 in Responding to Elder Abuse in GERiAtric Care - Provider questionnaire- REAGERA-P scale) than those who not entered

CONTACTS AND LOCATIONS:
Overall Officials: eman taha, Study Chair — Faculty of nursing, Alexandria university, Egypt
Locations (1):
- Alexandria university, Alexandria, Please Select A Country, Egypt

DOCUMENTS (1):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT06213025/Prot_000.pdf